CLINICAL TRIAL: NCT05631652
Title: Detection of Upper Gastrointestinal (GI) Bleeding Using a Novel Bleeding Sensor Capsule -Healthy Volunteers Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: EnteraSense Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CIP-019-02
Record Dates: First submitted 2022-11-14; First posted 2022-11-30 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Upper Gastrointestinal Bleeding
MeSH Terms: conditions — Gastrointestinal Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PillSense System (Experimental): All subjects were asked to swallow a PillSense Capsule, followed by the ingestion of autologous blood mixed with water, to verify the ability of the PillSense System to correctly identify blood.
  Interventions: Device: PillSense System

INTERVENTIONS:
Device: PillSense System — The device is composed of an orally ingested PillSense capsule and a wireless handheld PillSense receiver for real-time display of sensor data. The capsule contains an optical sensor for in-vivo detection of blood. The sensor capsule is used for diagnosis in patients with suspected acute bleeding in the upper gastrointestinal tract.

SUMMARY:
The objective of the investigation is to evaluate the feasibility of detecting blood in healthy volunteers after ingestion of autologous blood mixed with water.

DETAILED DESCRIPTION:
A total of 10 healthy volunteers were recruited to undergo a testing procedure. Subjects were instructed to ingest the PillSense Capsule with 100mL of water. The position of the capsule in the stomach was verified by fluoroscopy. Subjects were then asked to sequentially drink (every 5min) 2 mixtures containing 25mL of water and 25mL of their own blood obtained from a peripheral vein. The PillSense result ("blood detected" or " blood not detected") was recorded on Clinical Report Form after 5 minutes from capsule ingestion and after 5 minutes from the ingestion of both mixtures containing blood.

Subjects were followed-up for capsule passing.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 -60 years
2. Ability to give written informed consent

Exclusion Criteria:

1. Circulatory or hemodynamic instability with a clear need for urgent endoscopy or surgery (systolic blood pressure <100 mmHg,heart rate > 100 / min)
2. Known current stenosis of the GI tract
3. Presence of pacemaker or other implantable electronic device
4. Dysphagia or difficulties in swallowing pills the size of the capsule
5. History of achalasia or known esophageal dysmotility
6. History of gastroparesis
7. History of severe constipation (1 bowel movement per week or less)
8. Healthy volunteers who are currently pregnant or breastfeeding, or intend to become pregnant during the investigation
9. Active psychological issues preventing participation
10. Stomach bezoar
11. History of severe esophagitis
12. History of Crohn disease
13. History of diverticulitis
14. History of bowel obstruction
15. Suspected gastrointestinal tumor disease
16. Planned MRI investigation (MRI needed before the capsule is excreted)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2021-02-11 (Actual); Primary Completion 2021-03-11 (Actual); Study Completion 2021-03-11 (Actual)

PRIMARY OUTCOMES:
Device ability to detect the absence of blood | within 30 minutes
  Number of subjects in which PillSense capsule was able to identify the absence of blood post capsule ingestion and transmit the results to PillSense Receiver
Device ability to detect the presence of blood | within 30 minutes
  Number of subjects in which PillSense Capsule was able to identify the presence of blood post ingestion of a mixture containing autologous blood and transmit the results to PillSense Receiver

SECONDARY OUTCOMES:
Ability to ingest the capsule | within 30 minutes
  Number of subjects that were able to ingest the capsule
Absence of device-related adverse event | up to 4 weeks
  Number of subject that were able to naturally pass the capsule.
Absence of device-related adverse event | up to 4 weeks
  Number of subject that presented device-related adverse events (e.g. capsule retention, aspiration or bowel obstruction)

CONTACTS AND LOCATIONS:
Locations (1):
- Institut klinické a experimentální medicíny (IKEM),, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No